CLINICAL TRIAL: NCT00520416
Title: Prospective, Non-Randomized Evaluation of Carbon Dioxide Gas as a Contrast Agent in Comparison With Iodinated Contrast in Endovascular Aneurysm Repair
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: HS-06-00263
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Carbon Dioxide; Endovascular Abdominal Aortic Aneurym Repair; Prospective; Angiogram

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: There is no control or experimental group. The same patients undergoing endovascular AAA repair with serve as their own control
  Interventions: Procedure: Carbon dioxide angiogram

INTERVENTIONS:
Procedure: Carbon dioxide angiogram — see description of procedure

SUMMARY:
Endovascular repair of infrarenal abdominal aortic aneurysms (AAA) requires a contrast agent to identify the vascular anatomy and placement of the stent graft. Iodine contrast has traditionally been used, but has the potential to harm the kidneys. Another contrast agent is carbon dioxide gas. It has been proven safe to use, but the quality of the images it creates needs to be compared to iodine contrast. Patients in this study undergo the endovascular AAA repair as they normally, with the iodine contrast. At the end of surgery carbon dioxide gas contrast is given as an extra step. The images will be later evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infrarenal abdominal aortic aneurysm amendable to endovascular repair

Exclusion Criteria:

* renal failure or contraindication to receiving iodine contrast.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-10; Study Completion 2008-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred A Weaver, MD, Principal Investigator — University of Southern California
Locations (1):
- USC University Hospital, Los Angeles, California, United States